## Video Interventions for Dependence On Smoking (VIDeOS) for Cancer Patients: A Randomized Controlled Pilot Study

NCT number NCT06307496

Document Date 7/11/2024

## Consent Statement

You are being asked to volunteer for a research study. Research studies are voluntary and include only people who choose to take part. You are being asked to participate because you are a patient at MUSC with a cancer diagnosis who smokes. This is a research study to see if different materials about smoking cessation are helpful to people with cancer who want to quit smoking.

You will also be given a link to complete a survey online. The survey takes about 20 minutes to complete. After you complete this survey, you will be assigned to one of the study groups. Each group receives different resources about quitting smoking by text or email, depending on your preference. You will be assigned to a group based on random chance, like the flip of a coin. You will either receive an electronic version of a booklet to read or videos to watch whenever it is convenient for you during the next week.

You will be asked to complete additional 20 minute surveys one week, one month, and three months after you are assigned to a group and have a chance to review the resources. The surveys will ask you about your tobacco use, opinions about the materials, your cancer diagnosis, mood, and other things. You will also be asked to use a device (iCOquit) that measures your carbon monoxide levels. We will mail this device to you, and you will blow into the device to see how much carbon monoxide is in your body. We will ask you to enter the number into your one week, one month, and three month surveys. We will also ask for your name and email address in the surveys to allow us to send you a gift card code for participating. You will receive a \$25 Amazon gift code sent to your email for every survey you complete to compensate you for your time. You will receive a bonus \$25 gift code if you complete all surveys, for a total up to \$125. You can skip any question that you do not wish to answer. We will destroy identifiable information, including your name, phone number, and email address, when the study has been completed.

We will also conduct a brief chart review to get information about your cancer diagnosis and if you are receiving treatment. Once we obtain this information at the beginning of the study, we will not access your chart again.

If the materials used in the study prove to be effective, you may benefit from participating in this study, but that cannot be guaranteed. We will be asking you about your protected health information in this study, including about your cancer diagnosis. We will also be asking for your mailing address to send you your carbon monoxide detector and your email address to send you your gift card. Risks to participation include loss of confidentiality. Alternatives to participating in this study include choosing to not participate. Participating or choosing to not participate will not impact your healthcare at MUSC.

If you have additional questions, please contact the Study Primary Investigator.

Kinsey Pebley, PhD, MPH 843-779-5794 pebley@musc.edu

Are you interested in participating?

IRB Number: Pro00133913 Date Approved 7/11/2024

